CLINICAL TRIAL: NCT02009826
Title: Phase 0 Clinical Protocol: A Longitudinal and Multimodal Exploratory Study to Evaluate a Neuroinflammatory Hypothesis in Patients With Schizophrenia Compared to Young Healthy Subjects
Brief Title: Psychosis-Associated Neuroinflammation in Schizophrenia
Acronym: PANS
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other); Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, Dr Livia De Picker, Medical Doctor, Universiteit Antwerpen
Other Study IDs: CAPRI13/37/348; B300201318710 (Other: Belgian Study Registration Number)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Psychosis
Keywords: Schizophrenia; Psychosis; Neuroinflammation; Microglial activation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Neuroinflammatory Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy age- and sex-matched controls
  Interventions: Radiation: [18F]-PBR111 Positron Emission Tomography (PET); Behavioral: Cognitive and psychomotor tasks; Biological: Blood sampling
- Schizophrenia patients: Young schizophrenia patients 18-40y
  Interventions: Radiation: [18F]-PBR111 Positron Emission Tomography (PET); Behavioral: Cognitive and psychomotor tasks; Biological: Blood sampling

INTERVENTIONS:
Radiation: [18F]-PBR111 Positron Emission Tomography (PET) — [18F]-PBR111 radioligand to assess binding to TSPO
Behavioral: Cognitive and psychomotor tasks — Cognitive and psychomotor tasks on digitizing tablet
Biological: Blood sampling — Blood sampling for peripheral inflammatory and neurotoxicity markers

SUMMARY:
Previous research has suggested central nervous system inflammatory activity to be critically involved in disease development and progression in schizophrenia, with a complex interplay of inflammatory mechanisms leading to the development of brain abnormalities and medical symptoms related to schizophrenia. However, the mutual interactions of different inflammatory pathways and their relation to disease course have not been sufficiently studied. This study therefore aims to explore the interaction of neuroinflammatory mechanisms in patients with schizophrenia and to assess whether the inflammatory activity in schizophrenia is state-dependent and occurs mainly during psychotic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or woman between 18 and 40 years of age, inclusive.
* Have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in this study.
* Be medically stable on the basis of physical examination and vital signs performed at Screening.
* Be medically stable on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study.
* Be willing and able to adhere to the prohibitions and restrictions specified in the protocol.

Schizophrenia subjects:

* Fulfill DSM-V criteria for the schizophrenia spectrum (DSM-V #295.1-295.6, 295.9, 298.9)
* Be admitted to hospital for first-episode psychosis or acute relapse of psychosis, as defined by:

total score of ≥14 on the positive scale of the "Positive and Negative Syndrome Scale" (PANSS) and at least a score of 5 on 1 item or a score of 4 on 2 "psychotic" PANSS items P2, P3, P5 or G9 at Screening.

Exclusion Criteria:

* Use of nonsteroidal antiinflammatory drugs, paracetamol, immunosuppressant or immunostimulating drugs within 21 days of screening.
* Use of systemic corticosteroids within 21 days of screening.
* Has a history of drug or alcohol dependence according to DSM-V criteria, except nicotine or caffeine, within 6 months before screening.
* Has history of (co-morbid) somatization or mood disorder according to DSM-V criteria within 6 months before screening.
* Has a positive test result for drugs of abuse or for alcohol at screening or test day.
* Female subjects only: is pregnant or breastfeeding
* Has a history of chronic or acute physical illness associated with abnormal immune changes within the 2 weeks before the study.
* Leukocytosis (i.e., white blood cell count ≤ 11 x109 /L) on screening and test days.
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or HIV antibodies at screening.
* Has a medical history of any auto-immune disorder or chronic inflammatory disease.
* Has received electroconvulsive therapy in the last 6 months.
* Is currently enrolled in a study with an investigational study drug.
* Worsening or first time occurrence of significant suicidality
* Has donated blood within 3 months before screening.
* Has any condition that, in the opinion of the investigator, would compromise the wellbeing of the subject or the study or prevent the subject from meeting or performing study requirements.
* Low affinity binder of the TSPO, as determined by rs6971 polymorphism genotyping at Screening
* Use of benzodiazepines for 3x the half-life prior to PET-scan
* Presence of irremovable magnetic materials in or on the body
* Has a medical history of organic brain disease
* Has a medical history of traumatic brain injury
* Has a medical history of allergic reaction to any of the substances in the tracer fluid.
* Unwillingness or inability of subject to undergo PET and/or MRI scan (for example due to claustrophobia or lack of cooperation)

Healthy volunteers:

* Personal history of psychotic disorder
* Family history of psychotic or bipolar disorder in first-degree relatives
* Family history of auto-immune disorder in first-degree relatives

Schizophrenia patients:

- Calgary Depression Scale for Schizophrenia (CDSS) score >6 at screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young schizophrenia patients admitted to psychiatric hospital for acute relapse or first-episode of psychosis
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Regional VT of [18F]PBR111 | 2 years
  Regional distribution volume in tissue (VT) of 2-(6-chloro-2-(4-(3-fluoropropoxy)phenyl)imidazo(1,2-a)pyridin-3-yl)-N,N-diethylacetamide (PBR111) labelled with fluorine-18 (18F) in schizophrenia patients and age- , gender-, and translocator protein (TSPO) binding profile- matched healthy controls

SECONDARY OUTCOMES:
Peripheral markers | 2 years
  Levels and ratios of inflammatory and neurotoxicity markers in blood samples of schizophrenia patients compared to healthy age- and gender-matched healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Sabbe, MD PhD, Principal Investigator — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - Psychiatrisch Ziekenhuis Broeders Alexianen, Boechout, Antwerpen
  - Psychiatrisch Ziekenhuis St Norbertus, Duffel, Antwerpen
  - Psychiatrisch Ziekenhuis Sint-Amedeus, Mortsel, Antwerp